CLINICAL TRIAL: NCT00055198
Title: A Compassionate Use Protocol for Intravenous Daptomycin for the Treatment of Infections Due to Gram-Positive Bacteria That Cannot be Adequately Treated With Currently Available Therapy
Brief Title: Daptomycin for the Treatment of Infections Due to Gram-Positive Bacteria
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to low enrollment
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 3009-012; DAP-EAP-02-01 (Other: Cubist)
Record Dates: First submitted 2003-02-20; First posted 2003-02-21 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Gram-Positive Bacterial Infections
Keywords: Gram positive bacterial infections; expanded access program; resistant infections; bacteremia; Bacterial and fungal infections; bacterial infections
MeSH Terms: conditions — Gram-Positive Bacterial Infections; Bacteremia; Mycoses; Bacterial Infections | interventions — Daptomycin

INTERVENTIONS:
Drug: daptomycin

SUMMARY:
The purpose of this study is to provide daptomycin, an antibiotic, to patients who are failing conventional therapy, or who cannot take approved antibiotics for one reason or another.

ELIGIBILITY:
Main Inclusion Criteria:

* Infection caused by Staphylococcus aureus, Staphylococcus epidermidis, Enterococcus faecalis, or Enterococcus faecium that requires inpatient hospitalization and treatment with injectable antibiotics**
* Site of infection: complicated skin and skin structure infection; urinary tract infection; intra-abdominal infection; infective endocarditis; or bloodstream infection (including catheter-related).
* Pathogen resistant to, or patient intolerant of: beta-lactams, vancomycin, quinupristin/dalfopristin, or linezolid.
* Unable to receive any other standard commercially available antibacterial therapy for the infection.

Main Exclusion Criteria:

* Creatinine clearance less than 40 mL/min**
* Hemodialysis or peritoneal dialysis
* Admitted to the hospital for drug overdose or other conditions associated with rhabdomyolysis, or is expected to require repeated intramuscular injections
* Creatine phosphokinase (CPK) level greater than 2.5 times above the upper limit of normal (ULN) at screening; if the elevation in CPK can be attributed to an obvious cause (eg, surgery)**
* Central nervous system infection
* Pulmonary infection.

(**) An exemption may be granted for patients not satisfying these criteria following a conversation with the Medical Monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2002-12-19 (Actual); Primary Completion 2004-01-26 (Actual); Study Completion 2004-01-26 (Actual)